CLINICAL TRIAL: NCT04221867
Title: Feasibility and Therapeutic Potential of Free Fat Grafts in the Treatment of Esophageal Strictures
Brief Title: Feasibility and Therapeutic Potential of Free Fat Grafts in the Treatment of Esophageal Strictures (ESOGRAFT)
Acronym: ESOGRAFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hannes Kortekangas (Other Government)
Responsible Party: Sponsor-Investigator, Hannes Kortekangas, Gastrointestinal surgeon / Consultant in Division of Gastrointestinal Surgery, Turku University Hospital
Organization: Turku University Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESOGRAFT
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Esophageal Stricture; Fat Graft
Keywords: Esophageal Stricture; Fat Graft; Dilation
MeSH Terms: conditions — Esophageal Stenosis; Dilatation, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Esophageal stricture patients (Experimental): Patients suffering from benign esophageal stricture are treated with through-the scope CRE dilation balloon. Free fat graft is gathered from the abdominal subcutaneous fat. Fat graft is prepared and injected to the stricture site.
  Interventions: Procedure: Stricture dilation with CRE balloon; Procedure: Autologous fat grafting

INTERVENTIONS:
Procedure: Stricture dilation with CRE balloon — Esophageal stricture is treated by dilation therapy.
Procedure: Autologous fat grafting — Autologous fat graft is gathered and injected to stricture

SUMMARY:
In this study the investigators investigate the feasibility and therapeutic potential of free autologous fat grafting combined to dilation therapy in the treatment of benign esophageal strictures.

DETAILED DESCRIPTION:
In this study the investigators wish to proof the concept of free fat graft transfer into esophageal stricture via flexible video gastroscope.The investigators will recruit twenty patients suffering from (endoscopy proven) benign stricture of the esophagus. The Eckardt score is recorded upon recruitment and one day before operation.

The operation is performed at the gastroenterology outpatient clinic in Turku University Hospital by a gastrointestinal surgeon. The patient is sedated with alfentanil and midazolam. First, abdominal liposuction (roughly 20 ml) is performed under local infiltration anesthesia. The fat graft is processed into nano-fat using Tulip GEMS Single-Use NanoTransfer Set. Esophagoscopy with gastroscope is performed and stricture is visually graded (location, length, lumen) and photographed. Then esophageal stricture is biopsied with biopsy forceps and dilated with through-the-scope CRE(controlled radial expansion) balloon dilator. Prepared fat graft is injected beneath the mucosal layer at the stricture site (volume of 0,1-0,5 ml) at three locations. Patients are either discharged after two hours follow up or admitted to the inpatient ward, depending on the pre- and postoperative condition.

Patients are contacted by phone 1 week after the operation. Post-operative symptoms are recorded and patients are requested to contact the researcher if needed. Patient records are screened for pre- and postoperative symptoms, medication, long term illnesses and possible postoperative contacts to hospital.

Follow-up esophagoscopy is performed and biopsies taken three and 12 months after the first operation. The stricture site is visually graded and photographed. The Eckardt score is recorded. If the patient has problems with eating (Eckardt score dysphagia points more than 1) the stricture is re-dilated and fat grafting repeated.

If a patient would have recurrence in dysphagia before three months the patient is treated according to normal routine and dilation is repeated earlier.

The follow-up time is 12 months counting from the last fat grafting.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal stricture that has re-occurred at least once

Exclusion Criteria:

* Malignant etiology of esophageal stricture

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events at 3 months | 3 months
  Types, severity and probability of procedure related adverse events
Incidence of Treatment-Emergent Adverse Events at 12 months | 12 months
  Types, severity and probability of procedure related adverse events

SECONDARY OUTCOMES:
Change from Baseline Eckardt score at 3 months | 3 months
  Eckardt score is a validated symptom questionnaire used to measure achalasia symptoms. Esophageal stricture symptoms are similar to achalasia symptoms. Sub scales: Dysphagia, retrosternal pain, regurgitation, weight loss. Each sub scale 0-3 points. 0=none, 1=occasional / less than 5 kg, 2=daily / 5-10kg, 3= each meal /more than 10 kg. Total 0-12 points.
Change from Baseline Eckardt-score at 12 months | 12 months
  Eckardt score is a validated symptom questionnaire used to measure achalasia symptoms. Esophageal stricture symptoms are similar to achalasia symptoms. Sub scales: Dysphagia, retrosternal pain, regurgitation, weight loss. Each sub scale 0-3 points. 0=none, 1=occasional / less than 5 kg, 2=daily / 5-10kg, 3= each meal /more than 10 kg. Total 0-12 points.
Change from Baseline Stricture Lumen diameter at 3 months | 3 months
  Stricture photographed and lumen diameter measurement. Unit: closed biopsy forceps diameter.
Change from Baseline Stricture Lumen diameter at 12 months | 12 months
  Stricture photographed and lumen diameter measurement. Unit: closed biopsy forceps diameter.
Change from Baseline Stricture length at 3 months | 3 months
  Stricture length measured using shaft of biopsy forceps. Unit: mm.
Change from Baseline Stricture length at 12 months | 12 months
  Stricture length measured using shaft of biopsy forceps. Unit: mm.

CONTACTS AND LOCATIONS:
Overall Officials: Pauliina Hartiala, Surgeon, Study Director — Turku University Hospital